CLINICAL TRIAL: NCT02919514
Title: Effects of Physical Training on Hard, Sand and Soft Surfaces on Functional Ability and Incidence of Falls in Elderly With or Without History of Falls
Brief Title: Effect of Surfaces on Fall in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc.Prof.Dr., Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2561A10302245
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Falls, Accidental; Aging
Keywords: fall prevention; Aging; surfaces

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Physical training on hard surface (Active Comparator): Subject will participate in exercise training on a firm surface for 50 min/session, 3 days/week for 6 weeks in total.
  Interventions: Other: Physical training on sand surface.; Other: Physical training on soft surface.
- Physical training on sand surface (Experimental): Subject will participate in exercise training on a sand surface for 50 min/session, 3 days/week for 6 weeks in total.
  Interventions: Other: Physical training on hard surface.; Other: Physical training on soft surface.
- Physical training on soft surface (Experimental): Subject will participate in exercise training on a soft surface for 50 min/session, 3 days/week for 6 weeks in total.
  Interventions: Other: Physical training on hard surface.; Other: Physical training on sand surface.

INTERVENTIONS:
Other: Physical training on hard surface. — Physical training on hard surface.
  Arms: Physical training on sand surface; Physical training on soft surface
Other: Physical training on sand surface. — Physical training on sand surface.
  Arms: Physical training on hard surface; Physical training on soft surface
Other: Physical training on soft surface. — Physical training on soft surface.
  Arms: Physical training on hard surface; Physical training on sand surface

SUMMARY:
To investigate the effects of Thai dance exercises over 6 weeks on functional outcomes and incidence of fall in community-dwelling older individuals.

To compare effects of exercise training on hard, soft and sand surfaces in community-dwelling older individuals

ELIGIBILITY:
Inclusion Criteria:

* age at least 60 yr old
* fall

Exclusion Criteria:

* having pain (VAS >5)

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
10-meter walk test (10MWT) | 0,3 and 6 weeks
  The 10MWT quantifies walking speed that the results correlate to health status, morbidity rate and mortality rate; hence it has been suggested to be used as an important vital sign of elderly. Subjects walk along a 10meter walkway at a comfortable and fast gait speed. The time used over 4meters in the middle of the walkway will be recorded to minimize acceleration and deceleration effects. The average time required over the 3 trials will be converted to walking speed in m/s.

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, Ph.D., Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen, Thailand.
Locations (1):
- Khon Kaen University, Multiple Locations, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No